CLINICAL TRIAL: NCT02229032
Title: Genetic Analysis Between Charlotte's Web Responders Versus Non- Responders in a Dravet Population
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Denver Health Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0294
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Dravet Syndrome
Keywords: Dravet Syndrome; cannabidiol therapy; Charlotte's Web
MeSH Terms: conditions — Epilepsies, Myoclonic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — saliva for DNA analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dravet Sydrome: Patients with Dravet Syndrome who are self-seeking therapy with Charlotte's Web strain of medical marijuana with the assistance of a medical marijuana doctor, but are still naïve to therapy

SUMMARY:
There is tremendous curiosity about medical marijuana and the treatment of epilepsy. In a specific genetic epilepsy known as Dravet Syndrome, a mutation occurs affecting the SCN1A gene. A specific strain of marijuana known as Charlotte's Web, available in Colorado, may have activity in this catastrophic epilepsy syndrome. Anecdotal reports suggest both success and lack of response with this therapy. Genetic analysis of the differences between Dravet responders and non-responders may prove useful for identifying patients likely to be helped by this therapy, as well as shed light on the putative mechanisms by which marijuana may exert any antiepileptic effect.

ELIGIBILITY:
Inclusion Criteria:

* age 1-50 with gene confirmed Dravet Syndrome
* uncontrolled epilepsy, having failed at least 2 prior treatments (including appropriate Anti-epileptic drugs, ketogenic diet, vagus nerve stimulation Therapy)
* Seizure frequency should be more than 2 visually countable motor seizures per week (tonic clonic, tonic, clonic, myoclonic, or astatic)
* care providers able to identify convulsive seizures, drop attacks, or tonic seizures, or any combination of countable seizure types
* self- seeking therapy with Charlotte's Web strain of medical marijuana with the assistance of a medical marijuana doctor, but are still naïve to therapy
* care provider able to complete seizure count diary
* able to obtain oral swab sample from subject with Dravet Syndrome
* agree to forfeit any right to results of genetic analysis

Exclusion Criteria:

* subjects having non-epileptic seizures that are not distinguishable from epileptic seizures by the care provider
* prisoners
* pregnant women
* failure to forfeit right to results of genetic analysis

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Dravet Syndrome, ages 1-50, who are self- seeking therapy with Charlotte's Web strain of medical marijuana with the assistance of a medical marijuana doctor, but are still naïve to therapy
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
genetic differences between patients with Dravet Syndrome (SCN1A gene mutation) who appear to respond to high concentration cannabidiol (CBD) oil therapy versus those who do not. | 1 day
  Patients completing three months of therapy with a seizure reduction of >50% will be designated a "Responder" and patients who discontinue therapy for any reason prior to 3 months or have a <=50% seizure reduction will be designated "Non-Responder". Between-groups genetic analysis will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Edward Maa, MD, Principal Investigator — Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States